CLINICAL TRIAL: NCT00952263
Title: Open-Label, Dose Escalation Phase I Study in Healthy Volunteers to Evaluate the Safety and Pharmacokinetics of a Human Monoclonal Antibody (MBL-HCV1) Against Hepatitis C E2 Glycoprotein
Brief Title: Study in Healthy Volunteers to Evaluate a Human Monoclonal Antibody Against Hepatitis C
Acronym: MBL-HCV1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MassBiologics (Other)
Responsible Party: Deborah Molrine, MD, MassBiologics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-HCV1-09-01
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Hepatitis C; Phase I; Infusion; Pharmacokinetics; MBL-HCV1; Monoclonal antibody; Safety Assessment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBL-HCV1 (Experimental)
  Interventions: Biological: MBL-HCV1

INTERVENTIONS:
Biological: MBL-HCV1 — Single infusion of MBL-HCV1 at escalating doses as determined by cohort assignment: Cohort 1 @ 1 mg/kg, Cohort 2 @ 3 mg/kg, Cohort 3 @ 10 mg/kg, Cohort 4 @ 30 mg/kg, Cohort 5 @ 50 mg/kg.

SUMMARY:
This is a phase I, open-label, dose escalation study to evaluate the safety of MBL-HCV1 in healthy adult volunteers. Eligible volunteers will be admitted to a phase 1 unit for study infusion. A single dose of human monoclonal antibody will be administered. The study duration is 56 days. During this time, safety will be assessed via physical examinations, laboratory testing, concomitant medication usage and review of treatment emergent adverse events should they occur. Pharmacokinetics will be derived from analysis of blood samples obtained during the 56 day study.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose escalation study in healthy adult volunteers. Eligible volunteers will be admitted to a phase I unit for study infusion and be discharged after collection of a 24 hour post infusion sample. Thirty subjects are anticipated to be enrolled. There will be five cohorts of 6 subjects each. A single dose of human monoclonal antibody MBL-HCV1 will be administered on Day 0 and subjects will be followed for 56 days. Dose escalation to the next cohort will occur after review of safety data by the principal investigator, sponsor and an independent safety monitor through day 10 for all subjects in a cohort. Assessment of safety will be determined from vital sign measurements, physical examinations, hematology, chemistry and urinalysis laboratory testing, electrocardiograms, use of concomitant medications and review of treatment-emergent adverse events should they occur. Subjects will be evaluated at study visits on days 0, 1, 2, 3, 7, 14+/-1, 28+/-3 and 56+/-7. Blood samples and urinalysis for safety analyses will be drawn during screening and on days 0, 1, 3, 7 and 28+/-3. Blood samples for Pharmacokinetic analysis will be drawn on days 0, 1, 2, 3, 7, 14+/-1, 28+/-3 and 56+/-7. Blood samples for human anti-human antibody detection will be drawn on days 0, 14+/-1 and 56+/-7.

ELIGIBILITY:
Inclusion Criteria:

1. Study subject must have read, understood and provided written informed consent and HIPAA authorization after the nature of the study has been fully explained.
2. Be > or equal to 18 years of age and < or equal to 55 years of age.
3. Be in general good health without history of any of the conditions listed in exclusion criteria.
4. No use of any tobacco products for at least 6 months.
5. A woman must agree not to become pregnant from the time of study enrollment until at least 3 months after the completion of the monoclonal antibody infusion. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to use hormonal or barrier birth control with spermicidal gel.
6. Sexually active male subjects must use a barrier method of contraception during the course of the study.
7. Screening laboratory values must meet the following criteria:

   * WBC (>3,900 - <11,000/mm^3)
   * Platelets(>100,000/mm^3)
   * Hemoglobin (>10.5 gm/dl)
   * Creatinine (<1.1 x ULN)
   * BUN (<1.25 x ULN)
   * AST(<1.1 x ULN)
   * ALT (<1.1 x ULN)
   * Alkaline Phosphatase (<1.1 x ULN)
   * Bilirubin (<1.1 x ULN)
   * Glucose-nonfasting (>/=60 mg/dl and </=115 mg/dl)

Exclusion Criteria:

1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
2. Weight >90 kg
3. History of any of the following illnesses or conditions:

   * Cancer
   * Heart Disease
   * Diabetes mellitus
   * Respiratory condition (such as asthma requiring daily medication)
   * Autoimmune disorder
   * Blood dyscrasias
   * Psychiatric disorder that precludes compliance with protocol
   * Hepatitis
4. Any chronic condition requiring daily prescription or over-the-counter medicine except for vitamins and birth control products.
5. Drug or alcohol abuse within previous 12 months or a positive screen within 24 hours of monoclonal antibody administration.
6. History of a previous severe allergic reaction with generalized urticaria; angioedema or anaphylaxis.
7. Physical finding on examination considered clinically significant such as murmur (other than functional), hepatosplenomegaly, lymphadenopathy or focal neurological deficit.
8. Systolic blood pressure >140 or < 90 and/or diastolic blood pressure >90 on two separate readings.
9. Urinalysis positive for > trace protein, >5 rbc/hpf or >5 wbc/hpf
10. Positive serology for HIV antibody, HCV antibody or Hepatitis B surface antigen.
11. Positive urine pregnancy test during screening or within 24 hours of monoclonal antibody administration, or an unwillingness to undergo pregnancy testing.
12. Breast-feeding.
13. Receipt of licensed vaccine or other investigational study agent within previous 30 days.
14. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of escalating doses of a human monoclonal antibody against Hepatitis C E2 glycoprotein (MBL-HCV1) in healthy adults. | 56 days

SECONDARY OUTCOMES:
Determine pharmacokinetics of a human monoclonal antibody against Hepatitis C E2 glycoprotein (MBL-HCV1) given as a single intravenous infusion. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Swan, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States